CLINICAL TRIAL: NCT04276155
Title: Management of Anticoagulant Therapy Monitored by an Implantable Device With Telecardiology in Patients With Acute Coronary Syndrome Associated With de Novo Atrial Fibrillation Arrhythmia: A Prospective Multicenter Study
Brief Title: Management of Anticoagulant Therapy Monitored by an Implantable Device With Telecardiology in Patients With Acute Coronary Syndrome Associated With de Novo Atrial Fibrillation Arrhythmia
Acronym: SCA FA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHPAU2020/01
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation, Myocardial Infarction
Keywords: Acute Coronary Syndromes, Atrial Fibrillation, Anticoagulant therapy, Implantable device, Telecardiology.
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: prospective trial of therapeutic strategy, interventional, randomized and open-label, national and multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device (Experimental): Acute Coranary Syndrome and de novo Atrial Fibrilation patients treated by DAPT only, in association with an implantable cardiac monitoring device and a follow-up by telecardiology. The anticoagulant treatment will only be administered to patients presenting a recurrence of Atrial Fibrilation
  Interventions: Drug: non-systematic prescription of anticoagulant therapy
- Control (No Intervention): Acute Coranary Syndrome and de novo Atrial Fibrilation patients with standard management: DAPT in association with an anticoagulant treatment.

INTERVENTIONS:
Drug: non-systematic prescription of anticoagulant therapy — the prescription of anticoagulant is managed by an implantable device follow up
  Arms: Device

SUMMARY:
Patients with Acute Coronary Syndrome associated with de novo atrial fibrillation are randomized to benefit from either a conventional therapy associating dual antiplatelet therapy (DAPT) and anticoagulant or DAPT and an implantable monitoring device with a follow-up by telecardiology

DETAILED DESCRIPTION:
Acute Coronary Syndrome associated with de novo atrial fibrillation is not uncommon. It worsens the short-term, medium-term and long-term prognosis. It is then usual, according to ESC recommendations, to add to the DAPT, an anticoagulant treatment, which is a source of iatrogenic events, in particular hemorrhagic events. However, recurrence is not a certainty. Albeit variable, its highest rate is estimated to be 38%. Consequently, a well-conducted screening of atrial fibrillation recurrence could allow to treat only selected recurrent patients. At present, this screening can be carried out in a reliable and minimally invasive way with an implantable device with telecardiology. We propose a study for these patients with ACS associated with de novo AF. The study will be multicenter, randomized, open-label, with two arms: patient conventionally treated (DAPT + AC) and patient treated by DAPT + implantable device and followed for two years by telecardiology. This patient will only reintegrate the first arm in case of AF recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation diagnosed before hospitalization for acute coronary syndrome, whether treated or not.
* Atrial fibrillation still present at inclusion time.
* Transient atrial fibrillation due to a reversible disorder (thyrotoxycosis, pulmonary embolism, recent surgery).
* Acute coronary syndrome that has not been revascularized.
* Acute coronary syndrome surgically treated (bypass).
* Patient already on anticoagulant therapy.
* Scheduled aortocoronary bypass.
* Creatinine clearance < 30 ml per minute.

Exclusion Criteria:

Pathologic criteria :

* Atrial fibrillation diagnosed before hospitalization for acute coronary syndrome, whether treated or not.
* Atrial fibrillation still present at inclusion time.
* Transient atrial fibrillation due to a reversible disorder (thyrotoxycosis, pulmonary embolism, recent surgery).
* Acute coronary syndrome that has not been revascularized.
* Acute coronary syndrome surgically treated (bypass).
* Patient already on anticoagulant therapy.
* Scheduled aortocoronary bypass.
* Creatinine clearance < 30 ml per minute.

Bleeding risks :

* Contraindications to anticoagulant therapy.
* Active internal hemorrhage, clinically significant bleeding, bleeding non accessible to compression or bleeding diathesis within 30 days prior to selection visit.
* Platelet count < 90000/µL at the selection visit.
* Bleeding event in the twelve months prior to inclusion.
* Bleeding events detected either clinically or biologically (hemoglobinemia < 10g/dl).
* Elective surgery.

Comorbidities :

* Cardiogenic shock.
* Hyperthyroidism.
* Prior history of significant liver disease (acute hepatitis, active chronic hepatitis, cirrhosis) or liver function disorder detected at selection visit.
* Significant mitral valvular heart disease.

General :

* Patient under 18.
* Non menopausal woman or without contraception.
* Patient whose physical and / or mental health may have an impact on the compliance to the study.
* Participation in another biomedical research study (interventional or noninterventional) or participation in a research study within the 30 days prior to inclusion.
* Protected adults (under judicial protection, guardianship, or supervision).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of hemorrhagic events | 2 years
  To show that the introduction of an anticoagulant treatment in patients with ACS and de novo AF based on the data furnished by an implantable holter with remote monitoring is safer in terms of occurrence of hemorrhagic events than the systematic introduction of an anticoagulant treatment associated to DAPT based on the CHA2DS2-VASc score.
  CHA2DS2-Vasc score, derived from CHADS2 score. It assesses the risk of a person with atrial fibrillation (AF) without associated valve pathology, to experience an ischemic stroke, in other words, to assess the need for anticoagulant treatment. It ranges from 0 to 10. A score of 0 is considered a low risk. A score greater than or equal to 2 is considered a significant risk of embolic complication and should lead to discussion of the introduction of oral anticoagulant therapy.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Centre Hospitalier d'Aix en Provence, Aix-en-Provence
  - Centre hospitalier Chartres Louis Pasteur le Coudray, Chartres
  - Centre Hospitalier d'Haguenau, Haguenau
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Centre Hospitalier de Libournes, Libourne
  - Centre Hospitalier d'Annecy Genevois, Metz-Tessy
  - Centre hospitalier de Pau, Pau
  - Centre Hospitalier de Périgueux, Périgueux

IPD SHARING:
Plan to Share IPD: No